CLINICAL TRIAL: NCT04318145
Title: A Multi-Center, Unblinded, Single-Arm Study to Evaluate Sex Differences in the Acute Effects of PL-3994 on Myocardial cGMP Enhancement and Hemodynamics in Heart Failure With Preserved Ejection Fraction
Brief Title: Study to Evaluate Sex Differences in the Acute Effects of PL-3994 in Heart Failure Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study cancelled after Part A. Enrollment taking too long.
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL-3994-701
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure, Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — PL-3994

STUDY DESIGN:
Intervention Model Description: Part A: Single dose per subject, dose level ascension every 3 subjects. 5 dose levels are planned. An intermediate dose between planned doses may be chosen by the Sponsor/Investigator upon discussion after MTD is reached.
  Part B: Single dose, dose chosen from Part A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: PL-3994 Dose Ascension (Experimental): Dose ascension: up to 15 subjects with HFpEF. N = 3 per dose level, up to 5 dose levels.
  Interventions: Drug: PL-3994 Aqueous Intravenous Solution Dose Ascention
- Part B: PL-3994 Single Dose (Experimental): Up to 40 subjects with HFpEF (20 Females, 20 Males) will receive a single dose of PL-3994.
  Interventions: Drug: PL-3994 Aqueous Intravenous Solution Single Dose

INTERVENTIONS:
Drug: PL-3994 Aqueous Intravenous Solution Dose Ascention — Following appropriate dilution, PL-3994 will be injected intravenously by site personnel as a bolus dose followed by continuous infusion
  Other Names: PL-3994
  Arms: Part A: PL-3994 Dose Ascension
Drug: PL-3994 Aqueous Intravenous Solution Single Dose — Following appropriate dilution, PL-3994 will be injected intravenously by site personnel as a bolus dose followed by continuous infusion
  Other Names: PL-3994
  Arms: Part B: PL-3994 Single Dose

SUMMARY:
A Multi-Center, Unblinded, Single-Arm Study to Evaluate Sex Differences in the Acute Effects of PL-3994 on Myocardial cGMP Enhancement and Hemodynamics in Heart Failure with Preserved Ejection Fraction

DETAILED DESCRIPTION:
Multi-center, unblinded, dose ascending, two-part pilot study involving Part A, up to 15 subjects for dose ascension and optimization (N=3 per dose level, up to 5 dose levels) and Part B, 40 patients (n=20 women, n=20 men), with a single dose of PL-3994 after which hemodynamics will be measured by pulmonary artery catheter and pulmonary artery (mixed venous) and coronary sinus blood sampling will be performed to measure cGMP levels during a 15-minute observation period.

The objective of this study is to evaluate the acute effects of a single dose of intravenous PL-3994 on hemodynamics and myocardial cGMP expression.

The following endpoints will be assessed:

* Hemodynamics (including blood pressure, right atrial pressure, pulmonary artery pressure, pulmonary capillary wedge pressure, and cardiac output)
* Myocardial cGMP expression via coronary sinus sampling

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent.
2. Pre- or post-menopausal female or male age > 21 years
3. LVEF ≥ 45% by echocardiography within prior 6 months
4. Symptoms of HF requiring treatment with diuretics for ≥ 30 days prior to enrollment
5. Current symptoms of HF (NYHA class II-IV) at time of enrollment
6. 6. The subject has clinical indication for right heart catheterization for evaluation of HFpEF
7. Negative pregnancy test in a female of childbearing potential

Exclusion Criteria:

* A subject who meets ANY of the following exclusion criteria must not be enrolled.

  1. Orthostatic hypotension, systolic blood pressure <100 mm Hg, diastolic blood pressure < 50 mmHg.
  2. Any prior echocardiogram with LVEF < 40%
  3. Hemoglobin < 9 g/dl
  4. eGFR < 30 mL/min/1.73 m2
  5. Hemodynamically significant arrhythmias within prior 4 weeks
  6. Acute coronary syndrome, cardiac surgery, or percutaneous coronary intervention within prior 3 months
  7. Any of the following cardiac diagnoses: active myocarditis, hypertrophic cardiomyopathy, > moderate regurgitant valvular disease, any valvular stenosis, restrictive cardiomyopathy (including amyloid, sarcoid, or hemochromatosis), constrictive pericarditis, complex congenital heart disease, or pulmonary arterial hypertension
  8. Current need for IV inotropic medication
  9. Currently taking nitrates or having stopped nitrates within 24 hours of visit
  10. Currently taking antihistamines, antipsychotics, tri-cyclic antidepressants, catecholamines/related compounds, monoamine oxidase inhibitors, stimulants (including caffeine and nicotine), sympathomimetics, dopamine agonists. Additionally, medications that inhibit PDE activity will be prohibited during the study and for 5 half- lives prior to Day 1 so that cGMP measurements will not be affected
  11. Currently hospitalized for HF
  12. Any prior need for mechanical circulatory support
  13. Previous adverse reaction to the study drug
  14. Inability to comply with planned study procedures
  15. Pregnant or nursing mothers
  16. Participation in another study with an investigational drug or device within 30 days or a biologic study within 90 days prior to signing consent.
  17. Study participants must use method of birth control that has been approved by the Study Doctor and males must not donate sperm during the study and for 30 days after the last dose of study drug.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Part A: Dose Ascension | 1 day
  Reaching the maximum tolderated dose (MTD) as defined by meeting stopping criteria.
Part B: Coronary Sinus Levels | 1 day
  Coronary sinus levels of cGMP post PL-3994 infusion as compared to baseline.

SECONDARY OUTCOMES:
Part B: Blood pressure measured in mmHg | 1 day
  Measured at baseline (t=0) and at t=3, 6, 9, 12, and 15 minutes after the infusion of study drug.
Part B: Heart rate measured in beats per minute | 1 day
  Measured at baseline (t=0) and at t=3, 6, 9, 12, and 15 minutes after the infusion of study drug.
Part B: Right atrial pressure measured in mmHg | 1 day
  Measured at baseline (t=0) and at t=3, 6, 9, 12, and 15 minutes after the infusion of study drug.
Part B: Pulmonary artery pressure measured in mmHg | 1 day
  Measured at baseline (t=0) and at t=3, 6, 9, 12, and 15 minutes after the infusion of study drug.
Part B: Pulmonary capillary wedge pressure measured in mmHg | 1 day
  Measured at baseline (t=0) and at t=3, 6, 9, 12, and 15 minutes after the infusion of study drug.
Part B: Cardiac output measured in L/min. | 1 day
  Measured at baseline (t=0) and at t=3, 6, 9, 12, and 15 minutes after the infusion of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Sangiv J. Shah, MD, Principal Investigator — Northwestern University Medical Center
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No